CLINICAL TRIAL: NCT04076631
Title: A Prospective, Multicenter Clinical Study On Surgical Stages of Liver Cirrhosis In Patients With HBV-Related Hepatocellular Carcinoma
Brief Title: Surgical Stages of Liver Cirrhosis In Patients With Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: CXPJJH11900009
Record Dates: First submitted 2019-08-13; First posted 2019-09-03 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Surgically resected non-tumor liver tissues will be retained
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatocellular Carcinoma: Patients with hepatocellular carcinoma undergo open hepatectomy.

SUMMARY:
The investigators intend to perform a prospective, multicenter study to establish a set of clinical criteria for surgical stages of liver cirrhosis, which can be implemented to guide the surgical treatment of hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
HCC is the fifth most common malignancy in the world and ranks the third leading cause of tumor-related mortality. In China, more than 80% of HCC patients are accompanied by liver cirrhosis. Varied degrees of cirrhosis not only play an important role in selecting appropriate operative interventions for HCC patients, but are closely associated with tumor recurrence and long-term survival as well. Therefore, evaluating cirrhotic severity is essential for individualizing surgical modalities and predicting outcomes for patients with HCC. In recent years, investigators' group has proposed to stage the severity of liver cirrhosis through intraoperative liver morphological changes and preoperative cirrhotic severity scoring (TJ-CSS) model. Although the morphological classification of liver cirrhosis is of guiding significance for surgeons to determine the extent of hepatectomy, this method has some defects, such as subjectivity, lack of specific quantitative indicators and so on. Based on this, investigators propose to evaluate the severity of liver cirrhosis by measuring liver stiffness directly by Shaw hardmeter. Therefore, this prospective, multicenter clinical study intends to modify and perfect the preoperative cirrhotic severity scoring (TJ-CSS) and direct measurement of liver stiffness (DMS) grade established in the early period, so as to build a set of clinical standards for surgical liver cirrhosis classification, which can be used to guide the surgical treatment of HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 75 years of age, inclusive.
2. Patients who are clinically diagnosed as hepatocellular carcinoma and confirmed by postoperative pathology.
3. The liver function grade was Child-Pugh class A or class B, which can be restored to Child-Pugh class A within a short period of medical treatment.
4. Patients who undergo open surgery.
5. Patients have not been accompanied by serious physical diseases of heart, lung, brain, etc., and can generally tolerable for surgery.
6. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with tumors that oppress the main portal vein or main portal vein thrombus.
2. Patients that are accompanied with cavernous degeneration of portal vein.
3. Patients with hypersplenism caused by diseases of the blood system.
4. Patients suffer from serious acute and chronic diseases.
5. Patients with severe infectious diseases.
6. Patients with HIV-infectious or other AIDS-related disease.
7. Patients are drug abusers or have any psychological or mental conditions that potentially lead to poor study compliance.
8. Patients have any condition that in the judgement of the investigators would make the subject inappropriate for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo open liver resection with curative intent for HCC and meet the eligibility criteria from 6 hospitals in China (Wuhan Tongji Hospital, Wuhan Union Hospital, Wuhan Zhongnan hospital, Hubei Cancer Hospital, Shiyan Taihe Hospital, Xiangyang Central Hospital) will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Preoperative assessment of cirrhotic severity by cirrhotic severity scoring (TJ-CSS) | within 10 days prior to hepatectomy
  The calculation of TJ-CSS will be based on four clinical parameters (esophageal varices severity, portal vein diameter, spleen thickness and platelet account).
Liver stiffness measurement | during operation
  Liver stiffness will be measured by LX-C Shaw hardmeter.
Pathological stage of liver cirrhosis | Within 30 days after surgery
  Liver cirrhosis will be sub-staged according to Laennec staging system

SECONDARY OUTCOMES:
The effect of cirrhotic severity and extent of hepatectomy on the incidence of post-hepatectomy liver failure (PHLF) | postoperative day 5
  PHLF was diagnosed by the "50-50 criteria" characterized by the combination of a prothrombin time index of <50% and serum total bilirubin level of >50 mmol/L on postoperative day 5

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Liang BY, Zhang EL, Li J, Long X, Wang WQ, Zhang BX, Zhang ZW, Chen YF, Zhang WG, Mei B, Xiao ZY, Gu J, Zhang ZY, Xiang S, Dong HH, Zhang L, Zhu P, Cheng Q, Chen L, Zhang ZG, Zhang BH, Dong W, Liao XF, Yin T, Wu DD, Jiang B, Yuan YF, Zhang ZL, Chen YB, Li KY, Lau WY, Chen XP, Huang ZY. A combined pre- and intra-operative nomogram in evaluation of degrees of liver cirrhosis predicts post-hepatectomy liver failure: a multicenter prospective study. Hepatobiliary Surg Nutr. 2024 Apr 3;13(2):198-213. doi: 10.21037/hbsn-22-410. Epub 2023 Mar 15. PMID 38617471